CLINICAL TRIAL: NCT02424812
Title: Evaluation Of The Unilever Lifebuoy School-Based Handwashing Campaign (School Of 5) In Rural Bihar, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Hindustan Unilever Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ciff001
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Diarrhea
Keywords: handwashing; behavior
MeSH Terms: conditions — Diarrhea; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): school based handwashing education programme
  Interventions: Behavioral: Lifebuoy School of Five Handwashing Intervention
- Control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Lifebuoy School of Five Handwashing Intervention
  Arms: Intervention

SUMMARY:
The effect of large scale handwashing and hygiene promotion campaigns on handwashing behaviour, diarrhoea and respiratory infections is not known. While Intensive small scale interventions have achieved improvements in handwashing behaviour and reductions in diarrhoea and respiratory infections, it is not clear whether realistic and scalable interventions delivered across large areas achieve effects large enough to be of public health interest. The Unilever "School of 5" Lifebuoy campaign is such a scalable intervention that is being rolled out across the state of Bihar during 2015 to 2017. The proposed study aims at evaluation the effect of this campaign on handwashing behaviour in school aged children and their mothers, and on diarrhoea and respiratory infections in the same children and their younger siblings.

DETAILED DESCRIPTION:
The Unilever Lifebuoy School-Based Handwashing campaign ("School of 5") aims at raising hygiene awareness and the importance of handwashing with soap among school children and their parents attending rural Indian schools. The campaign is funded by Unilever Ltd India and Children's Investment Fund Foundation (CIFF). CIFF is paying for this evaluation. The aim of this trial is to evaluate the effect of the Unilever Lifebuoy School-Based Handwashing campaign on 1) handwashing behaviour in school aged children and their mothers/carers (primary outcome), 2) psychosocial indicators of hygiene behaviour in the target population; 3) on diarrhoea in children under 5 years of age living in families with school children attending intervention schools.

We will conduct a cluster randomised trial (CRT) of 320 villages in one district of Bihar State, India. The unit of treatment allocation will be villages, as some villages have more than one school. We expect selection of 320 villages to result in about 400 eligible schools. Schools are eligible to receive the intervention if they have more than 150 children enrolled in the school register. 160 villages will be randomised to receive the intervention at the beginning of the study before assessing the study outcomes ("intervention schools/villages") and 160 will be randomised to receive the intervention at the end of the programme after completing all research activities ("control schools/villages").

The research activities will be done in four phases. Phase 1 will be a conducted before the intervention within a subset of 20 villages of the total population of randomised study villages (10 intervention - 10 control), randomly selected from two blocks (administrative units at sub-district level) in the district. The aim is to obtain a baseline measurement of handwashing habits using the sticker diary methodology developed by Unilever.

In Phase 2 we will evaluate the impact of the intervention on handwashing behaviour in the target population, i.e. handwashing at specified times in school children and their mothers. Hygiene behaviour will be measured by two methods: 1) sticker diary (measured by revisiting the Phase 1 villages and households); 2) Direct structured observation of handwashing. For the structured observation study we will recruit households from 12 control and 12 intervention villages that are different from the phase 1 villages. We will further evaluate the early effect of the intervention on knowledge of intervention content, attitudes and motivations related to hygiene behaviour and handwashing in school children and their parents. The results of phase 2 will tell us whether the intervention changed the target behaviours as a basis for achieving any health impact. Based on the results of Phase 2 we will make the following decisions for Phase 3 in collaboration with the co-funder (CIFF): 1) if Phase 2 indicates a marked behaviour change with the potential to impact on health, we will proceed with the measurement of the main health outcomes in all study villages. 2) If there is no major behaviour change potentially impacting on health, we will focus on the process documentation, qualitative research and with the aim of obtaining knowledge for improving the current campaign and increase our learning from the programme.

Upon completion of Phase 3, or phase 2 if no phase 3 is conducted, we will conduct a final handwashing behaviour change assessment (Phase 4) in the study area in the phase 2 villages, and in a further district in Bihar to assess the impact of the intervention on handwashing behaviour across a wider area, and the sustainability of the changes. This phase will use the same methods as in Phase 2, and also include an economic evaluation of the programme.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled households have a child that attends a school in the village that has more than 150 children on the school register.
* Enrolled households further have a child under 5 years.

Exclusion Criteria:

* none of the above

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2628 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Handwashing with soap | 3 months after intervention, single contact
  handwashing behaviour will be assessed by direct (structured) observation by a female field observer. Specifically, observers will identify 3 occasions of handwashing (before eating, after toilet use, and after child care). The primary outcome of the study will be the proportion of these observed occasions at which the subject washed hands with soap. The outcome will be observed in school children and adult household members.

SECONDARY OUTCOMES:
Diarrhoea | 6 months to 9 months post intervention
  Diarrhoea will be assessed as the 2 week period prevalence of diarrhoea in children under 5 years. Diarrhoea will be defined as 3 or more loose stools on at least one day at any time during the past 2 weeks if the loose stools were associated with general signs of being unwell: unwilling to play, abdominal pain, vomiting, treatment sought. The symptoms will be assessed by the use of questionnaires administered to the primary carer of the child.

CONTACTS AND LOCATIONS:
Overall Officials: Wolf-Peter Schmidt, PhD, MD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- KAAPRO, Patna, Bihar, India

IPD SHARING:
Plan to Share IPD: No